CLINICAL TRIAL: NCT00600015
Title: A Randomized Double-Blind Placebo-Controlled Phase II Trial of Sorafenib and Erlotinib or Erlotinib Alone in Previously Treated Advanced Non-Small Cell Lung Cancer
Brief Title: Sorafenib/Erlotinib Versus Erlotinib Alone in Previously Treated Advanced Non-Small-Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SCRI LUN 160
Record Dates: First submitted 2007-12-26; First posted 2008-01-24 (Estimated); Results first posted 2012-09-21 (Estimated); Last update posted 2022-03-10 (Actual); Status verified 2022-02

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer; Advanced; Sorafenib; Erlotinib; Double-blind; Placebo-controlled
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Sorafenib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Combination Therapy (Experimental): Erlotinib + Sorafenib
  Interventions: Drug: Erlotinib + Sorafenib
- Placebo (Placebo Comparator): Erlotinib + Placebo
  Interventions: Drug: Erlotinib + Placebo

INTERVENTIONS:
Drug: Erlotinib + Sorafenib — Patients who are randomized to Cohort A will take sorafenib 400 mg (2 x 200-mg tablets) orally twice a day, and erlotinib 150 mg orally once a day.
  Other Names: Tarceva; Nexavar
  Arms: Combination Therapy
Drug: Erlotinib + Placebo — Patients who are randomized to Cohort B will take erlotinib 150 mg orally once a day and placebo orally twice a day.
  Other Names: Tarceva
  Arms: Placebo

SUMMARY:
This trial will investigate the use of the newer targeted agents erlotinib and sorafenib in patients with stage IIIB or stage IV NSCLC who have received 1-2 prior chemotherapy regimens. Patients will be randomized to receive erlotinib (150 mg/day) and sorafenib (400 mg twice daily), or erlotinib (150 mg/day) and a placebo.

DETAILED DESCRIPTION:
The rationale of this study is to combine two distinct kinase inhibitors to evaluate synergistic inhibition of angiogenesis and epidermal growth factor receptor (EGFR) signaling. Erlotinib is a oral tyrosine kinase inhibitor that targets EGFR. Sorafenib is a oral tyrosine kinase inhibitor targeting vascular endothelial growth factor receptor (VEGFR), platelet derived growth factor receptor beta, Raf-1, Flt-3, and C-kit. These agents also do not exhibit overlapping adverse event profiles which provided additional support for studying this combination therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed locally advanced or metastatic NSCLC (unresectable stage IIIB or stage IV). Eligible histologies include adenocarcinoma and squamous cell carcinoma. Patients with recurrent disease after treatment for localized NSCLC are also eligible. Cytologic specimens obtained by brushings, washings, or needle aspiration are acceptable.
* At least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques, or as >= 10 mm with spiral computerized tomography (CT) scan according to the Response Evaluation Criteria in Solid Tumors (RECIST).
* Failure of at least one, and no more than two prior cytotoxic chemotherapy regimens for advanced disease (either due to progressive disease or toxicity).
* Recovery from any toxic effects of prior therapy to <= grade 1.
* Completion of radiation therapy at least 28 days prior to the start of study treatment (not including palliative local radiation). Previously irradiated lesions in the advanced setting cannot be included as target lesions unless clear tumor progression has been observed since the end of radiation.
* An ECOG performance status of 0-2.
* Absolute neutrophil count (ANC) >= 1,500, platelets >= 75,000.
* Hemoglobin >= 9 g/dL (within 7 days prior to study treatment).
* International normalized ratio (INR) <= 1.5 or prothrombin time (PT)/partial thromboplastin time (PTT) within normal limits (WNL) of the institution
* Serum creatinine <= 1.5 x institutional upper limit of normal (ULN) within 7 days prior to study treatment.
* Transaminases <= 3 x institutional ULN
* Agreement of female patients of childbearing potential and male patients who have partners of childbearing potential to use an effective form of contraception to prevent pregnancy during treatment, and for a minimum of 90 days thereafter.
* Patients who have treated brain metastases >= 4 weeks out (with surgery and/or radiation therapy) and no evidence of CNS progression.

Exclusion Criteria:

* Past or current history of neoplasm (other than the entry diagnosis), with the exception of treated non-melanoma skin cancer or carcinoma in-situ of the cervix, or other cancers cured by local therapy alone, and a disease-free survival (DFS) >= 3 years.
* Patients who have mixed tumors with small-cell elements are ineligible.
* Pregnancy or lactation.
* Prior treatment with EGFR TKIs or VEGFR TKIs for NSCLC. [NOTE: prior cetuximab and/or bevacizumab use is permitted].
* Significant cardiac disease within 90 days of starting study treatment
* Myocardial infarction within 6 months prior to initiation of study treatment.
* Cardiomegaly on chest imaging or ventricular hypertrophy on electrocardiogram (ECG)
* Poorly controlled hypertension
* Unstable angina (anginal symptoms at rest).
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy.
* Presence of cardiac disease that, in the opinion of the investigator, increases the risk of ventricular arrhythmia.
* A serious underlying medical condition that would impair the ability of the patient to receive protocol treatment.
* A major surgical procedure, open biopsy, or significant traumatic injury within 28 days of beginning treatment, or anticipation of the need for major surgery during the course of the study.
* Stroke or transient ischemic attack (TIA) within the past 6 months.
* Any prior history of hypertensive crisis or hypertensive encephalopathy.
* Pulmonary hemorrhage/bleeding event >= grade 2 within 28 days of study treatment.
* Any other non-pulmonary hemorrhage/bleeding event >= grade 3 within 28 days of study treatment.
* Evidence or history of bleeding diathesis or coagulopathy.
* Serious non-healing wound, ulcer, or bone fracture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2008-02; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Spigel, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (16):
- United States (16):
  - Florida Cancer Specialists, Fort Myers, Florida
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Wellstar Cancer Research, Marietta, Georgia
  - Kansas City Cancer Centers, Overland Park, Kansas
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Methodist Cancer Center, Omaha, Nebraska
  - Cancer Care of Western North Carolina, Asheville, North Carolina
  - Oncology Hematology Care, Cincinnati, Ohio
  - Mid Ohio Oncology/Hematology, Inc./ The Mark H. Zangmeister Center, Columbus, Ohio
  - South Carolina Oncology Associates, PA, Columbia, South Carolina
  - Chattanooga Oncology Hematology Associates, Chattanooga, Tennessee
  - Family Cancer Center, Collierville, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Coastal Bend Cancer Center, Corpus Christi, Texas
  - Virginia Cancer Institute, Richmond, Virginia

REFERENCES:
- [Background] Spigel DR, Burris HA 3rd, Greco FA, Shipley DL, Friedman EK, Waterhouse DM, Whorf RC, Mitchell RB, Daniel DB, Zangmeister J, Bass JD, Hainsworth JD. Randomized, double-blind, placebo-controlled, phase II trial of sorafenib and erlotinib or erlotinib alone in previously treated advanced non-small-cell lung cancer. J Clin Oncol. 2011 Jun 20;29(18):2582-9. doi: 10.1200/JCO.2010.30.7678. Epub 2011 May 16. PMID 21576636

RESULTS

PARTICIPANT FLOW:
Groups:
- Combination Therapy: sorafenib (400 mg orally twice a day) plus erlotinib (150 mg orally daily)
- Placebo: Placebo twice daily orally plus erlotinib (150 mg orally daily)
Period: Overall Study
Arm/Group | Combination Therapy | Placebo
Started | 111 | 55
Completed | 51 (Completed >=2 cycles) | 20 (Completed >=2 cycles)
Not Completed | 60 | 35

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Combination Therapy | Placebo | Total
Number analyzed (Participants) | 111 | 55 | 166
Age, Continuous [Median (Full Range); unit: years] | 65 [44 to 88] | 65 [45 to 83] | 65 [44 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 29 | 78
  Male | 62 | 26 | 88
Region of Enrollment [Number; unit: participants]
  United States | 111 | 55 | 166

OUTCOME MEASURES:

1. Primary Outcome: Overall Objective Response Rate (ORR)
Description: Overall response rate (ORR) is defined as the percentage of patients who have a partial or complete response to therapy. Responses were assessed by the Response Evaluation Criteria in Solid Tumors (RECIST; version 1.0).
  Complete Response: Disappearance of all target lesions, and disappearance of all non-target lesions.
  Partial Response: At least a 30% decrease in the sum of the longest diameter of target lesions (taking as reference the baseline sum of longest diameters)
Time Frame: 18 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Combination Therapy | Placebo
Number analyzed (Participants) | 111 | 55
percentage of participants | 8.1 [3.77 to 14.83] | 10.9 [4.11 to 22.25]

2. Primary Outcome: Progression Free Survival (PFS)
Description: Progression-free survival is defined as the time from the first day of treatment until the day tumor progression was documented. Response was evaluated using the Response Evaluation Criteria in Solid Tumors (RECIST).
  Progressive Disease (PD): Appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions
Time Frame: 18 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Combination Therapy | Placebo
Number analyzed (Participants) | 111 | 55
Months | 3.38 [2.30 to 3.81] | 1.94 [1.77 to 3.65]

3. Primary Outcome: Disease Control Rate (DCR)
Description: Disease Control Rate (DCR) is defined as the percentage of patients who have a partial/complete/stable response to therapy. Responses were assessed by the Response Evaluation Criteria in Solid Tumors (RECIST; version 1.0).
  Complete Response: Disappearance of all target lesions, and disappearance of all non-target lesions.
  Partial Response: At least a 30% decrease in the sum of the longest diameter of target lesions (taking as reference the baseline sum of longest diameters) Stable Response: Neither sufficient shrinkage to qualify for partial response, nor sufficient increase to qualify for progressive disease (taking as reference the smallest sum of diameters since the treatment started).
Time Frame: 18 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Combination Therapy | Placebo
Number analyzed (Participants) | 111 | 55
percentage of participants | 54 [44 to 64] | 38 [25 to 52]

4. Secondary Outcome: Duration of Response
Description: Duration of response is defined as the time from when objective response is realized until time to first documented disease progression. Disease progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. Objective Response = CR + PR. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI or CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions.
Time Frame: 18 months
Measure: Mean (Standard Error); unit: months
Arm/Group | Combination Therapy | Placebo
Number analyzed (Participants) | 111 | 55
months | 4.6430 (1.0048) | 5.2234 (0.4571)

5. Secondary Outcome: 6-month PFS
Description: Progression free survival is defined as the time from the first day of treatment until the day tumor progression was documented. Response was evaluated using the Response Evaluation Criteria in Solid Tumors (RECIST). Progressive Disease (PD): Appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions (1). Percentage of participants who were progression free at 6 month from the start of treatment is reported here.
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Combination Therapy | Placebo
Number analyzed (Participants) | 111 | 55
percentage of participants | 29 | 22

6. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the first treatment until date of death due to any cause. In the absence of confirmation of death or lack of data beyond follow-up period, the survival time was censored to last date the participant was known to be alive.
Time Frame: 18 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Combination Therapy | Placebo
Number analyzed (Participants) | 111 | 55
Months | 7.62 [5.35 to 10.54] | 7.23 [4.04 to 12.58]

ADVERSE EVENTS:
Groups:
- All Study Participants: Reported SAEs and AEs for all study participants -
  Combination Therapy: Erlotinib + Sorafenib Placebo: Erlotinib + Placebo
Arm/Group | All Study Participants
Serious Adverse Events (participants affected / at risk) | 77/166
Other Adverse Events (participants affected / at risk) | 141/166
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Study Participants (N=166)
Hemorrhage (Blood and lymphatic system disorders) | 1 (1)
Cardiopulmonary Arrest (Cardiac disorders) | 4 (4)
Supraventricular Arrhythmia - Atrial Fibrillation (Cardiac disorders) | 1 (1)
Supraventricular Arrhythmia - Atrial Tachycardia (Cardiac disorders) | 2 (2)
Supraventricular Arrhythmia (Cardiac disorders) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 1 (2)
Cardiac Troponin I (Cardiac disorders) | 1 (1)
Chest Pain (Nervous system disorders) | 1 (1)
Death (General disorders) | 2 (2)
Dehydration (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Obstruction - Small Bowel (Gastrointestinal disorders) | 1 (2)
Fistula - Esophagus (Gastrointestinal disorders) | 1 (1)
Perforation - Small Bowel (Gastrointestinal disorders) | 1 (1)
Enteritis (Gastrointestinal disorders) | 2 (2) — Diverticulitis
Esophagitis (Gastrointestinal disorders) | 1 (1) — GERD
Vomiting (Gastrointestinal disorders) | 1 (1)
Obstruction - Esophagus (Gastrointestinal disorders) | 1 (1)
Liver Dysfunction (Hepatobiliary disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Pneumonia (Infections and infestations) | 4 (6)
Sepsis (Infections and infestations) | 1 (1)
Fungal Infection (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Failure To Thrive (Metabolism and nutrition disorders) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Weakness (Musculoskeletal and connective tissue disorders) | 2 (3)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal - Other (Musculoskeletal and connective tissue disorders) | 1 (1) — Diskitis
Progressive Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 18 (18)
Pain (Nervous system disorders) | 9 (10)
Neurology - Other (Nervous system disorders) | 1 (1) — Neurodeficit
Seizure (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Mental Status (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
CNS Ischemia (Nervous system disorders) | 1 (1) — CVA
Cystitis (Renal and urinary disorders) | 1 (1) — Hematuria
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 14 (16)
ARDS (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Adult Respiratory Distress Syndrome
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Airway Obstruction - COPD (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Thrombosis/Thrombis/Embolism (Vascular disorders) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Study Participants (N=166)
Anemia (Blood and lymphatic system disorders) | 141 (141)
Leukopenia (Blood and lymphatic system disorders) | 24 (24)
Neutropenia (Blood and lymphatic system disorders) | 15 (15)
Thrombocytopenia (Blood and lymphatic system disorders) | 37 (37)
Diarrhea (Gastrointestinal disorders) | 121 (121)
Anorexia (Gastrointestinal disorders) | 84 (84)
Rash (Skin and subcutaneous tissue disorders) | 109 (109)
Hand-Foot (Skin and subcutaneous tissue disorders) | 43 (43)
Fatigue (General disorders) | 120 (120)
Hypertension (Cardiac disorders) | 25 (25)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites.